CLINICAL TRIAL: NCT07130708
Title: Advancing Humanitarian Healthcare: Exploring the Potential of Robotic Telesurgery in Remote Settings - A Multicentric Prospective Study
Brief Title: Exploring the Potential of Robotic Telesurgery in Remote Settings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Principal Investigator, Vipul Patel, MD, Medical Director, AdventHealth Cancer Institute Urologic Oncology Program Medical Director, AdventhHealth Celebration Global Robotics Institute, AdventHealth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2294288
Record Dates: First submitted 2025-06-18; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-06

CONDITIONS: Prostate Carcinoma; Prostate Disease
Keywords: Robotic Prostatectomy; Prostate Cancer; Telesurgery
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Exploring the Potential of Robotic Telesurgery in Remote Settings (Experimental): Telesurgery
  Interventions: Device: Telesurgery utilizing Microport Medbot Robotic Platform

INTERVENTIONS:
Device: Telesurgery utilizing Microport Medbot Robotic Platform — A robotic surgery for prostate disease via telesurgery, where a highly trained surgeon performs the operation remotely using a secure internet connection.

SUMMARY:
This study involves a type of robotic surgery called telesurgery, where a highly trained surgeon performs the surgical procedure using a secure internet connection to operate on a patient in a different location. Urologists from The goal of this study is to find out how safe and effective telesurgery is when used in real hospitals. The study aims to understand how well Telesurgery works in different settings, what technical challenges might come up (like internet speed or delays), and how it can be used to train new surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 90
* Male or female
* Eligible participants for this telesurgery study must have a clearly defined indication for robotic urologic surgery, specifically:

  * Localized Prostate Cancer (ICD-10: C61), appropriate for robotic radical prostatectomy.

OR

-Benign Prostate diseases appropriate for robotic simple prostatectomy (ICD-10: N40) These diagnoses are confirmed by clinical examination, imaging, and/or pathology prior to surgical planning. Patients with vague or unspecified urologic conditions will be excluded to ensure the safety and appropriateness of the surgical intervention.

* Primary diagnosis of urinary system disease and prostate disorders (C61 and N40.1) scheduled to undergo treatment with robotic surgery. These patients don't have access to robotic surgery in their routine and the study will give them the opportunity to have advanced technology and the gold-standard treatment with experts in the field.
* Willing to participate in the study
* Mentally capable of comprehending the study protocol

Exclusion Criteria:

* Patients who, based on multidisciplinary evaluation (surgical, anesthetic, and medical), are deemed not suitable for robotic surgery due to high perioperative risk. This includes but is not limited to:

  * Uncontrolled cardiovascular, pulmonary, or metabolic disease.
  * Severe anesthetic risk classified as ASA Class IV or higher.
* Patients enrolled in another interventional research study that may interfere with surgical safety or outcomes.
* Patients unwilling or unable to comply with the perioperative and follow-up schedule.
* Vulnerable populations are excluded from this study, including:

  * Minors (under 18 years old)
  * Prisoners
  * Cognitively impaired or decisional incapacitated individuals

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2025-06-14 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2033-07-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measures (Endpoints) | The measured time frame for this outcome will be measured by the investigator and tech team from the start of the surgical procedure through the stop time of the surgical procedure. Approximately 90 minutes in length.
  One of the investigator's primary outcome measures is the safety and feasibility of the Microport Medbot Robotic Platform for use in Telesurgery through maintaining a stable connection. The investigator will monitor feasibility through perioperative connectivity assessment provided by the platform.
  Outcome of Latency- Medbot platform measures in milliseconds. This is monitored by the investigator. Measured in Milliseconds per round trip time (ms/RTT). The acceptable threshold is under 200ms.
  Robotic Platform Performance Logs- The robotic system itself continuously logs and reports performance metrics, including latency.
  Dedicated Tech team: Oversees and monitors connection status throughout procedure.
Secondary Endpoints | This will be measured by the investigator from the start of the surgical procedure through the completion of the surgical procedure.
  Investigators assessment of and response to perioperative complications (complications observed will be classified using the Clavien-Dindo Classification with Grades I thru V).
Safety and Feasibility: Maintenance of stable connection | The measured time frame for this outcome will be measured by the investigator and tech team from the start of the surgical procedure through the stop time of the surgical procedure. Approximately 90 minutes in length.
  One of the investigator's primary outcome measures is the safety and feasibility of the Microport Medbot Robotic Platform for use in Telesurgery through maintaining a stable connection. The investigator will monitor feasibility through perioperative connectivity
  Outcome: Bandwidth and Network Stability- The surgical team monitors bandwidth to ensure a consistent, high-speed internet connection. Bandwidth measured in megabits per second (Mbps). The goal of 100Mbps is recommended.
  Measurement is made through tracking on data transmission rates reported by the robotic system itself which continuously logs and reports data in real time.
  Dedicated Tech Team: Oversees and monitors connection status throughout the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- AdventHealth, Celebration, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
We plan to publish multiple articles during the study, using the full de-identified dataset from all patients or focusing on specific subsets of the data to highlight particular types of surgeries or groups of procedures.

REFERENCES:
- [Background] Rocco B, Moschovas MC, Saikali S, Gaia G, Patel V, Sighinolfi MC. Insights from telesurgery expert conference on recent clinical experience and current status of remote surgery. J Robot Surg. 2024 Jun 4;18(1):240. doi: 10.1007/s11701-024-01984-w. PMID 38833111
- [Background] Reddy SK, Saikali S, Gamal A, Moschovas MC, Rogers T, Dohler M, Marescaux J, Patel V. Telesurgery: A Systematic Literature Review and Future Directions. Ann Surg. 2025 Aug 1;282(2):219-227. doi: 10.1097/SLA.0000000000006570. Epub 2024 Oct 22. PMID 39435556
- [Background] Patel V, Dohler M, Marescaux J, Saikali S, Gamal A, Reddy S, Rogers T, Patel E, Oliva R, Satava R, Moschovas MC. Expanding Surgical Frontiers Across the Pacific Ocean: Insights from the First Telesurgery Procedures Connecting Orlando with Shanghai in Animal Models. Eur Urol Open Sci. 2024 Oct 21;70:70-78. doi: 10.1016/j.euros.2024.09.009. eCollection 2024 Dec. PMID 39502103
- [Background] Dohler M, Saikali S, Gamal A, Moschovas MC, Patel V. The crucial role of 5G, 6G, and fiber in robotic telesurgery. J Robot Surg. 2024 Nov 16;19(1):4. doi: 10.1007/s11701-024-02164-6. PMID 39549181
- [Background] Moschovas MC, Saikali S, Dohler M, Patel E, Rogers T, Gamal A, Marquinez J, Patel V. Advancing Telesurgery Connectivity Between North and South America: the first Remote Surgery Conducted Between Orlando and Sao Paulo in Animal Models. Int Braz J Urol. 2025 Jan-Feb;51(1):e20240601. doi: 10.1590/S1677-5538.IBJU.2024.0601. No abstract available. PMID 39556854
- [Background] Patel V, Moschovas MC, Marescaux J, Satava R, Dasgupta P, Dohler M. Telesurgery collaborative community working group: insights about the current telesurgery scenario. J Robot Surg. 2024 May 31;18(1):232. doi: 10.1007/s11701-024-01995-7. No abstract available. PMID 38819496
- [Background] Patel V, Marescaux J, Covas Moschovas M. The Humanitarian Impact of Telesurgery and Remote Surgery in Global Medicine. Eur Urol. 2024 Aug;86(2):88-89. doi: 10.1016/j.eururo.2024.04.029. Epub 2024 May 18. PMID 38762391